CLINICAL TRIAL: NCT00864266
Title: Biological Factors Predicting Response to Chemotherapy in Advanced Non Small Cell Lung Cancer : a Prospective Study
Brief Title: Biological Factors Predicting Response to Chemotherapy in Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Lung Cancer Working Party (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 01082
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: Non small cell lung carcinoma; Chemotherapy; Response prediction
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): After obtaining the biopsy, patients will be treated by standard chemotherapy (the regimen has to be in agreement with the ELCWP guidelines, available on the website www.elcwp.org)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Standard cisplatin-based chemotherapy in agreement with the ELCWP guidelines (available on the website www.elcwp.org)

SUMMARY:
The primary aim of the study is to identify a predictive molecular signature for response to chemotherapy, according to WHO criteria, in patients with non-small cell lung cancer by studying the transcriptome (miRNAs and mRNAs) and the single nucleotide polymorphism (SNPs) by using high throughput techniques.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of non-small-cell lung cancer (NSCLC)
* Obtention of a biopsy of the tumour according to the procedure defined in the protocol
* NSCLC of any stage to be treated by standard conventional first-line chemotherapy, as defined in the ELCWP guidelines (www.elcwp.org)
* Presence of at least one assessable lesion
* Availability for participating in the detailed follow-up of the protocol
* Signed informed consent.
* Age above 18 years

Exclusion Criteria:

* Patient who was previously treated with chemotherapy for NSCLC or who has any contra-indication precluding the administration of conventional chemotherapy for NSCLC
* NSCLC treated by exclusive surgery or radiotherapy
* A history of prior malignant tumour, except non-melanoma skin cancer or in situ carcinoma of the cervix or of the bladder or cured malignant tumour (more than 5-year disease free interval)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-03 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Response rate | response will be assessed every 3 cycles of chemotherapy according to WHO criteria

SECONDARY OUTCOMES:
Survival | Survival will be dated from the date of treatment
Progression-free survival | Period between the date of treatment and the date of first progression or death
Duration of response | period between the day of treatment and the date of first progression in patients with an objective response

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Berghmans, MD, Study Chair — European Lung Cancer Working Party
Locations (6):
- Belgium (6):
  - Department of Pneumology Clinique Saint-Luc, Bouge
  - Department of Intensive Care Unit and Thoracic Oncology Institut Jules Bordet, Brussels
  - Service de Pneumologie Hôpital Erasme, Brussels
  - Department of Pneumology Hôpital Saint-Joseph, Gilly
  - Hôpital Ambroise Paré, Mons
  - Department of Pneumology Centre Hospitalier de Mouscron, Mouscron

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Berghmans T, Ameye L, Lafitte JJ, Colinet B, Cortot A, CsToth I, Holbrechts S, Lecomte J, Mascaux C, Meert AP, Paesmans M, Richez M, Scherpereel A, Tulippe C, Willems L, Dernies T, Leclercq N, Sculier JP; European Lung Cancer Working Party. Prospective Validation Obtained in a Similar Group of Patients and with Similar High Throughput Biological Tests Failed to Confirm Signatures for Prediction of Response to Chemotherapy and Survival in Advanced NSCLC: A Prospective Study from the European Lung Cancer Working Party. Front Oncol. 2015 Jan 28;4:386. doi: 10.3389/fonc.2014.00386. eCollection 2014. PMID 25674536
- [Derived] Berghmans T, Ameye L, Willems L, Paesmans M, Mascaux C, Lafitte JJ, Meert AP, Scherpereel A, Cortot AB, Cstoth I, Dernies T, Toussaint L, Leclercq N, Sculier JP; European Lung Cancer Working Party. Identification of microRNA-based signatures for response and survival for non-small cell lung cancer treated with cisplatin-vinorelbine A ELCWP prospective study. Lung Cancer. 2013 Nov;82(2):340-5. doi: 10.1016/j.lungcan.2013.07.020. Epub 2013 Aug 7. PMID 24007627
- See also: (Click here for more information on the protocol) — http://www.elcwp.org